CLINICAL TRIAL: NCT06007599
Title: Surgical Wound Healing With and Without the Use of Skin Adhesive in Primary TKA
Brief Title: Wound Healing in Primary TKA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MAUS2023-2092
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Total Knee Replacement; Wound Complication

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: suture with skin adhesive (Active Comparator): After surgery the closure technique utilized by the surgeons will be subcuticular running 3-0 monocryl sutures without skin adhesive
  Interventions: Procedure: Skin closure using skin adhesive
- Group B: suture without skin adhesive (Active Comparator): After surgery the closure technique utilized by the surgeons will be subcuticular running 3-0 monocryl sutures with skin adhesive.
  Interventions: Procedure: Skin closure without skin adhesive

INTERVENTIONS:
Procedure: Skin closure using skin adhesive — Wound closure using subcuticular running 3-0 monocryl sutures with skin adhesive
  Arms: Group A: suture with skin adhesive
Procedure: Skin closure without skin adhesive — Wound closure using subcuticular running 3-0 monocryl sutures without skin adhesive
  Arms: Group B: suture without skin adhesive

SUMMARY:
Wound complications after total knee arthroplasty (TKA) can arise from many patient-specific factors, such as vascular or immune-related medical conditions, obesity, and smoking, among others. The development of early wound complications can lead to increased length of hospital stay and more serious complications, including deep infection and major subsequent surgery. However, there are modifiable variables that could affect the risk of getting wound complications, such as the closure technique. This study aims to analyze the difference in rates of wound complications using two different closure techniques in primary TKA.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old that will undergo primary TKA with a midline approach

Exclusion Criteria:

* Previous knee arthroplasty surgeries or midline scars
* TKA secondary to oncologic or traumatic etiologies
* BMI ≥ 40
* uncontrolled diabetes (measured by a Hgb A1c above 8)
* reported allergy to skin adhesive
* immunodeficiencies
* bleeding disorders
* anticoagulation other than ASA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
wound complications | 90 days
  Assessed using Photographic documentation of the wound
Patient satisfaction | 90 days
  Assessed using the POSAS (patient and observer scar assessment scale) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States